CLINICAL TRIAL: NCT06228690
Title: Comparison of Gold Fish Exercises and Cervico-thoracic Postural Correction Training in Patients With Temporo-mandibular Joint Dysfunction
Brief Title: Comparison of Gold Fish Exercises and Cervico-thoracic Postural Correction Training in Patients With TMJD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S22C08G30024
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Temporomandibular Joint; Temporomandibular Joint Dysfunction
Keywords: Temporomandibular joint dysfunction.; Gold Fish exercises; Cervico-thoracic postural correction training
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gold Fish exercises (Experimental): Gold Fish exercises for the flexibility of TMJ that will target the Jaw muscles.
  Interventions: Other: Gold Fish exercises
- Cervico-thoracic postural correction training. (Experimental): Cervico-thoracic postural correction training for upper thoracic and neck muscles.
  Interventions: Other: Cervico-thoracic postural correction training
- Conventional PT treatment (Active Comparator): Conventional PT including Hot Pack for 10mins, Active-Passive neck Stretching Exercise + jaw Isometric Exercises.
  Interventions: Other: Conventional PT treatment

INTERVENTIONS:
Other: Gold Fish exercises — Specific exercise for the flexibility of TMJ that will target the Jaw muscles. Frequency: 3 times/week for 4 weeks Intensity: moderate intensity (pain free) Time: 30-45 minutes Type: Gold Fish exercises for jaw flexibility, pain and maximum mouth opening.
  Arms: Gold Fish exercises
Other: Cervico-thoracic postural correction training — Cervico-thoracic postural correction training for upper thoracic and neck muscles.
  Frequency: 3 times/week for 4 weeks Intensity: moderate intensity (pain free) Time: 30-45 minutes Type: Muscle energy technique to improve range of motion, pain and maximum mouth opening.
  Arms: Cervico-thoracic postural correction training.
Other: Conventional PT treatment — Conventional PT including Hot Pack for 10mins, Active-Passive neck Stretching Exercise + jaw Isometric Exercises.
  * Frequency: hold followed by 5secs rest. 2-3times for 3 times/week for 4 weeks, Intensity: moderate-high intensity (depending on pain tolerance) Time: 30-45 mins for Active-Passive neck Stretching.
  * Frequency: 3secs hold, 6 times repetitions for Isometric Exercises. Type: conventional treatment for pain, ROM, MMO.
  Arms: Conventional PT treatment

SUMMARY:
The aim of this randomized controlled trial is to determine the effect of Gold Fish exercises and cervico-thoracic postural correction training in patients with temporo-mandibular joint dysfunction to improve pain, ROM and maximum mouth opening of jaw.

DETAILED DESCRIPTION:
Goldfish Exercise works on the principle of pulsatile motion of Goldfish in water & thereby imitating the same motion for health benefits. It can be thought of stretching the fibrous bands, reducing TMJ stiffness & resulting in improvement of mouth opening. It would be beneficial to use this technique on daily basis and as far there are no contraindications of this exercise because it's done within the pain limits & further progression depends on the mouth opening of the patient.

Posture can affect the three-dimensional movement of the jaw during opening which is seen most clearly in the slumped posture as reduced maximal mouth opening. While mouth opening and head extension are linked, there is variability in the amount of head extension when opening wide and the relationship between head extension and mouth opening is negated when opening in a slumped posture. This has implications for the association of neck dysfunction, posture, and temporo-mandibular joint disorder which should be explored further.

ELIGIBILITY:
Inclusion Criteria:

- Age group 20-40 Both males and females Forward head posture and temporo-mandibular joint dysfunction for more than 3 months.

Pain provocation during neck movement, chewing and yawning; more than 5 on the Visual analogue scale.

Exclusion Criteria:

* History of cervical spine injury or surgery
* Pain due to underlying condition i.e. neoplasm, vascular disease
* Infection, inflammation
* Erupting 3rd molar/dental origin
* Congenital condition of cervical spine or TMJ

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-08-03 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Vernier calipers | 4 weeks
  The maximum mouth opening distance is a generally accepted measurement to estimate temporomandibular joint mobility and function. The maximum distance is measured from the incisal edge of the maxillary central incisors to the incisal edge of the mandibular central incisors at the midline. The value is measured in millimeters.
: visual analogue scale | 4 weeks
  VAS is a qualitative pain measurement tool that assigns integer numbers between zero and 10 to different pain levels, where zero means no pain and 10 means excruciating pain. VAS is a reliable scale to measure jaw pain.
Inclinometer | 4 weeks
  It is an instrument that measures the available range of motion at a joint.
Neck disability index | 4 weeks
  It is used for disability in patients related to any musculoskeletal neck condition. Total score is presented in percentage. A higher score tells greater disability while 0 means no disability.
Temporomandibular Dysfunction Disability Index (TDI) | 4 weeks
  The TMJ Disability Index questionnaire focuses on determining prior and post treatment level of function and patient's quality of life and what aspects are affected and to what degree. A total score out of 40 was calculated and converted into percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Dentovilla Esthetic and Medical Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No